CLINICAL TRIAL: NCT06233409
Title: A Novel Sandwich Technique of Minimally Invasive Keratoplasty for Corneal Perforation
Acronym: STMIK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: zhangyi2023
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Corneal Perforation, Corneal Stromal Lenticule,Sandwich Technique
Keywords: Corneal perforation, Corneal stromal lenticule,Sandwich technique
MeSH Terms: conditions — Corneal Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lenticules group: Morphology of cornea and intra-ocular pressure were obtained by optical coherence tomography, Non-contact tonometer, Slit-lamp photography
- Penetrating keratoplasty group: Morphology of cornea and intra-ocular pressure were obtained by optical coherence tomography, Non-contact tonometer, Slit-lamp photography

SUMMARY:
The goal of this type of study to describe a new sandwich technique of minimally invasive keratoplasty (STMIK) by using SMILE-extracted lenticules for treatment corneal perforation and effectiveness.

The main question[s] it aims to answer are: 1.Corneal perforations require urgent attendances for prompt treatments. How can we restore the integrity of the eyeball as soon as possible, reduce complications, and restore vision in the case of lack of corneal material according to the conditions that may be obtained.

2.In China, nearly 1 million lenticules are obtained through all-femtosecond surgery every year. How to reuse and turn waste into precious materials for clinical application is an important study.

Participants will understand and signed the informed consent to take this new method for the treatment of their corneal perforations disease, which will obtain good results, but there may be a certain risk of complications.The main tasks participants will be asked to cooperate as required.The clinical eye check includes the test of includes visual acuity, slit lamp, anterior segment phase, anterior segment OCT and IOP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with corneal perforation who are willing to undergo treatment with this new technique;
2. The size of cornea perforation was ≦ 3mm

Exclusion Criteria:

1. The size of cornea perforation was >3mm
2. Patients with corneal perforation who were unwilling to be treated with this new technique.
3. Patients who could not be followed up regularly.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients premedicated for keratoplasty surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
A Novel Sandwich Technique for Corneal Perforation | one year
  By sandwiching the corneal lenticules interlamellar implantation, STMIK as an alternative novel treatment and effective procedure that provides an option to restore the corneal integrity and improve vision in patients with corneal perforations.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided